CLINICAL TRIAL: NCT05578391
Title: PHASE II Clinical Trial Randomized And Controlled To Assess Need Of Oxygen On Day 14 After Administration Of Passive Immunotherapy In Patients Infected By SARS-CoV-2 With Risks Factors For Severe Disease
Brief Title: Passive Immunotherapy In Patients With SARS CoV-2
Acronym: CoV-PlasGal
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fundacin Biomedica Galicia Sur (Other)
Collaborators: Health Knowledge Agency (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CoV-PlasGal
Record Dates: First submitted 2022-09-17; First posted 2022-10-13 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Convalescent plasma (Experimental)
  Interventions: Biological: Convalescent plasma
- Conventional treatment (No Intervention)

INTERVENTIONS:
Biological: Convalescent plasma — Admistration of one unit of convalescent plasma
  Arms: Convalescent plasma

SUMMARY:
Plasma from convalescent individuals (convalescent plasma, CP) has been used for more than a hundred years for the treatment of infectious diseases. Among patients with COVID-19, it has been used first, in patients with severe infection. Although it is a safe treatment, it has not been possible to demonstrate a reduction in mortality in cases of acute respiratory distress syndrome.

The objective of the clinical trial is to evaluate the efficacy and safety of the early use (less than 5 days of symptoms) of CP in patients infected with SARS-CoV-2 with risk factors for severe disease.

The primary efficacy endpoint was the proportion of patients requiring oxygen therapy to maintain saturation >93% on day 14. Secondary objectives included, evaluation of the safety of the treatment, measured as the appearance of some adverse event related to the CP infusion; the evolution of COVID-19 symptoms and WHO progression scale status at day 14 and 28 after inclusion; the need for hospitalization due to progression of COVID-19. COVID-19 progression was considered as worsening of respiratory symptoms requiring oxygen therapy at some point. Finally, death from any cause was evaluated at 28 days, after inclusion in the study.

ELIGIBILITY:
Inclusion Criteria:

Patients with SARS-CoV-2 infection, confirmed by any validated microbiological technique, and with one or more symptoms associated with COVID-19 with ≤5 days of evolution and with an oxygen saturation ≥93% breathing room air.

In addition, the patients had to present some risk factor for severe disease:

* Chronic heart failure (NYHA ≥ 2)
* Arterial hypertension under pharmacological treatment
* Chronic lung disease: COPD (bronchitis, emphysema or chronic obstruction) with dyspnoea at least on moderate exertion, or moderate-severe asthma (that required inhaled corticosteroids to control symptoms or had received systemic corticosteroids during the last year due to decompensation)
* Chronic renal failure (glomerular filtration rate <60 ml/min/1.73 m², by CKD- ILD)
* Diabetes mellitus requiring pharmacological treatment or obesity grade ≥ I (BMI ≥30 Kg/m2).
* Patients ≥65 years were included, regardless of other risk factors.

Exclusion Criteria:

* Duration of symptoms >5 days
* Dyspnoea at rest
* Need for supplemental oxygen to maintain O2 saturation >93%
* Solid neoplastic or haematologic disease (except skin cancer) with active treatment in the last 3 months before the onset of symptoms
* Patients under chronic corticosteroid treatment (equivalent to prednisone 10 mg/d for at least 28 days) or immunosuppressive treatment
* Decompensated liver cirrhosis
* Participation in another clinical trial
* History of hypersensitivity to haematological derivatives
* Pregnancy or lactation,
* AST/ALT >5 times the upper limit of normal or at baseline in patients with chronic liver disease
* Any condition that in the opinion of the investigator limits participation in the study.
* Patients who had received monoclonal antibodies against SARS-CoV-2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Requirement for oxygen therapy to maintain saturation >93% | Day 14
  Proportion of patients that need oxygen to achieve a saturation >93%

SECONDARY OUTCOMES:
Safety of the treatment with CP | Day 1
  Safety of CP treatment was evaluated by the appearance of any adverse event related to the infusion
Evolution of COVID-19 symptoms | Day 14 and 28
  Proportion of patients with 1+2 WHO progression scale. This scale was developed by a special World Health Organization (WHO) committee for quantifying COVID-19 illness severity.
  1. = Not hospitalized without limitation in activity (no symptoms)
  2. = Not hospitalized with limitation in activity (continued symptoms)
  3. = Hospitalized not on supplemental oxygen
  4. = Hospitalized on supplemental oxygen by mask or nasal prongs
  5. = Hospitalized on non-invasive ventilation or high flow nasal cannula
  6. = Hospitalized, intubated and mechanically ventilated
  7. = Hospitalized, intubated, mechanically ventilated and requiring additional organ support (pressors, renal replacement therapy)
  8. = Death
Requirement for hospitalization due to worsening of symptoms | Until day 28
  Worsening of symptoms was evaluated using the WHO progression scale
  1. = Not hospitalized without limitation in activity (no symptoms)
  2. = Not hospitalized with limitation in activity (continued symptoms)
  3. = Hospitalized not on supplemental oxygen
  4. = Hospitalized on supplemental oxygen by mask or nasal prongs
  5. = Hospitalized on non-invasive ventilation or high flow nasal cannula
  6. = Hospitalized, intubated and mechanically ventilated
  7. = Hospitalized, intubated, mechanically ventilated and requiring additional organ support (pressors, renal replacement therapy)
  8. = Death

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Álvaro Cunqueiro, Vigo, Spain

IPD SHARING:
Plan to Share IPD: No